CLINICAL TRIAL: NCT03294343
Title: Risk-Reducing Surgeries of Salpingo-oophorectomy With/Without Hysterectomy for Carriers With Mutation Genes of Hereditary Ovarian Cancer
Brief Title: Risk-Reducing Surgeries for Hereditary Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SOHHO
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis; Ovariectomy; Hysterectomy
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome; Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — Salpingo-oophorectomy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HBOCS (Experimental): For carriers with mutation genes of BRCA1, BRCA2 (both belonging to mutation genes of hereditary breast and ovarian cancer syndrome, HBOCS) and ATM, BRIP1, RAD51, RAD51C, and RAD51D (all belonging to mutation genes of other hereditary ovarian cancer syndrome), if they demand for risk-reducing surgeries, counseling, decision-making analysis, then salpingo-oophorectomy only by laparoscopy and long-term follow-up are provided.
  Interventions: Procedure: salpingo-oophorectomy only by laparoscopy
- Lynch syndromes (Experimental): for carriers with mutation genes of MLH1, MSH2, MSH6, PMS2, EPCAM (all belonging to mutation genes of Lynch syndromes) and STK11, , if they demand for risk-reducing surgeries, counseling, decision-making analysis, then salpingo-oophorectomy with hysterectomy by laparoscopy and long-term follow-up are provided.
  Interventions: Procedure: salpingo-oophorectomy with hysterectomy by laparoscopy
- Refusal to surgery (Other): For carriers with any mutation genes (BRCA1, BRCA2, ATM, BRIP1, RAD51, RAD51C, RAD51D, STK11, MLH1, MSH2, MSH6, PMS2 and EPCAM) but refusal to any risk-reducing surgeries, counseling, decision-making analysis, and then long-term follow-up are provided.
  Interventions: Other: Follow-up

INTERVENTIONS:
Procedure: salpingo-oophorectomy only by laparoscopy — Salpingo-oophorectomy are provided for carriers with mutation genes of BRCA1, BRCA2 (both belonging to mutation genes of hereditary breast and ovarian cancer syndrome, HBOCS) and ATM, BRIP1, RAD51, RAD51C, and RAD51D (all belonging to mutation genes of other hereditary ovarian cancer syndrome). Detailed multi-disciplinary counseling, decision-making analysis before surgeries, and long-term follow-up and health management after surgeries are provided for all participants.
  Arms: HBOCS
Procedure: salpingo-oophorectomy with hysterectomy by laparoscopy — Salpingo-oophorectomy with hysterectomy are provided for carriers with mutation genes of MLH1, MSH2, MSH6, PMS2, EPCAM (all belonging to mutation genes of Lynch syndromes) and STK11. Detailed multi-disciplinary counseling, decision-making analysis before surgeries, and long-term follow-up and health management after surgeries are provided for all participants.
  Arms: Lynch syndromes
Other: Follow-up — Detailed multi-disciplinary counseling, decision-making analysis and long-term follow-up are provided for carriers with any mutation genes but refusal to any risk-reducing gynecologic surgeries
  Arms: Refusal to surgery

SUMMARY:
Based on studies of "Inherited Susceptible Genes Among Epithelial Ovarian Cancer" (NCT03015376, clinicaltrials.gov) and "Cohort Study of Universal Screening for Lynch Syndrome in Chinese Patients of Endometrial Cancer" (NCT03291106, clinicaltrials.gov), we provide risk-reducing surgeries of salpingo-oophorectomy with/without hysterectomy for healthy carriers with mutation genes of hereditary ovarian cancer, which is defined ovarian cancer with relevant pathogenic mutations.

ELIGIBILITY:
Inclusion Criteria:

* Carriers with known and definite mutation genes of hereditary ovarian cancer.
* With children and without further requirement of pregnancy.
* No less than 35 years for carriers with mutation gene of BRCA1.
* No less than 40 years for carriers with mutation gene of BRCA2.
* No less than 45 years for carriers with mutation genes of BRIP1, RAD51C, RAD51D and RAD51.
* No less than 50 years for carriers with mutation genes of ATM, MSH2, MLH1, SH6, PMS2, EPCAM and STK11.

Exclusion Criteria:

* Without children.
* Not reaching appreciate ages.
* With contraindications of laparoscopy.
* Refusal of risk-reducing surgeries.

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Occult cancer or precancerous lesion in histological specimen | 5 years
  Precancerous lesions include serous tubal intraepithelial carcinoma (STIC) and endometrial intraepithelial neoplasia (EIN)

SECONDARY OUTCOMES:
Overall survival | 10 years
  Duration from surgery to death
Incidence of primary peritoneal carcinoma | 10 years
  Incidence of primary peritoneal carcinoma after reception or refusal risk-reducing salpingo-oophorectomy
Incidence of primary uterine cancer | 10 years
  Incidence of primary uterine cancer after reception or refusal risk-reducing hysterectomy

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, China/Beiing, China

IPD SHARING:
Plan to Share IPD: Undecided